CLINICAL TRIAL: NCT02669355
Title: Observational Study to Determine the Effect of Wearing of White Coat on Patient Satisfaction in Indian Out Patient Department (OPD) Setting
Brief Title: Effect of Wearing of White Coat on Patient Satisfaction in Indian Out Patient Department (OPD) Setting
Status: Completed | Type: Observational
Sponsor: Columbia Asia (Other)
Responsible Party: Principal Investigator, Dr.Sharath Kumar, Rheumatology Consultant, Columbia Asia
Other Study IDs: IEC/2015/RP/17
Record Dates: First submitted 2015-10-28; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Patient Compliance; Physician-Patient Relations
Keywords: White coat physician attire
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Doctor's attire acts as an important criteria in setting up good relationship between patient and physician. Recent evidence as well as strong viewpoints have highlighted the possible harm of wearing a white coat. In order to get the patient's perspective on the same, this observational study is being conducted to determine the effect of wearing a white coat on patient satisfaction in an Indian setting , in patients who visit rheumatology outpatient department,in Columbia Asia Hospitals,Bangalore,India.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged equal to or greater than 18 years, attending the rheumatology OPD in Columbia Asia Hospitals,Bangalore.

Exclusion Criteria:

* Patient who have come only for diagnostic or therapeutic procedure or for second opinion.
* Patients without plan for follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged above 18 years who come to consult in Rheumatalogy OPD in all three Columbia Asia Hospitals situated in Bangalore are taken into study.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in patient satisfaction scores (if any) between patients visiting a rheumatologist for the first time based on the whether the physician dons an apron or not. | 50 days

SECONDARY OUTCOMES:
Change in rate of compliance with medications between patients visiting a rheumatologist for the first time based on the whether the physician dons an apron or not. | 3 weeks to 1 month.
Change in rate of compliance with follow up visits (if any) between patients visiting a rheumatologist for the first time based on the whether the physician dons an apron or not. | 3 weeks to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sharath Kumar, MBBS,MD,DNB, Principal Investigator — Columbia Asia Hospitals,Bangalore
Locations (1):
- Columbia Asia Hospitals, Bangalore, Karnataka, India

REFERENCES:
- [Background] Petrilli CM, Mack M, Petrilli JJ, Hickner A, Saint S, Chopra V. Understanding the role of physician attire on patient perceptions: a systematic review of the literature--targeting attire to improve likelihood of rapport (TAILOR) investigators. BMJ Open. 2015 Jan 19;5(1):e006578. doi: 10.1136/bmjopen-2014-006578. PMID 25600254
- [Background] Hughes LD, Done J, Young A. A 5 item version of the Compliance Questionnaire for Rheumatology (CQR5) successfully identifies low adherence to DMARDs. BMC Musculoskelet Disord. 2013 Oct 8;14:286. doi: 10.1186/1471-2474-14-286. PMID 24103582
- [Background] de Klerk E, van der Heijde D, Landewe R, van der Tempel H, van der Linden S. The compliance-questionnaire-rheumatology compared with electronic medication event monitoring: a validation study. J Rheumatol. 2003 Nov;30(11):2469-75. PMID 14677194
- [Background] Fernandes E. Doctors and medical students in India should stop wearing white coats. BMJ. 2015 Jul 21;351:h3855. doi: 10.1136/bmj.h3855. No abstract available. PMID 26198987
- See also: Original feedback form of the General Medical Council of the UK (United Kingdom)which has been modified for this study — http://www.gmc-uk.org/doctors/revalidation/colleague_patient_feedback_resources.asp